CLINICAL TRIAL: NCT05607862
Title: Effects of a Home-based Therapeutic Exercise Program on Frailty in Patients With Parkinson's Disease
Brief Title: Home Physiotherapy in Frailty in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, María Cruz Sousa Fraguas, Principal Investigator. Physiotherapist., University of Oviedo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-398 Parkinson´s disease.
Record Dates: First submitted 2022-10-30; First posted 2022-11-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease; Physical Therapy Modalities; Frailty
Keywords: Home physiotherapy
MeSH Terms: conditions — Parkinson Disease; Frailty | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will continue with its usual medical-pharmacological treatment, and will also receive a multi-component exercise program and health education guidelines.
  Interventions: Other: Home Physiotherapy Group
- Control Group (Other): The control group will be given health education guidelines and will continue with their usual medical-pharmacological treatment.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Home Physiotherapy Group — The intervention group will receive 2 sessions per week for 8 weeks supervised and assisted by a physiotherapist at the patient's home. Muscle strengthening exercises of the lower and upper limbs, stretching, coordination and balance exercises, gait re-education with the relevant technical aids, a pattern of exercises to be performed daily by the patient and health education guidelines will be carried out.
  Arms: Intervention Group
Other: Control Group — The control group will be given health education guidelines and will continue with their usual medical-pharmacological treatment. All patients included in this study will receive physiotherapy treatment, and those in the control group will be treated once the intervention and the post-intervention assessment have been completed.
  Arms: Control Group

SUMMARY:
The aim of this protocol is to evaluate the effects of a home-based therapeutic exercise program applied in patients with PD to reverse frailty. The design of this study is experimental, prospective, randomized and single blind. The study population that will be part of this study will be men and women with a diagnosis of PD belonging to the Health Area V of the Health Service of the Principality of Asturias, Spain.

DETAILED DESCRIPTION:
Introduction: Parkinson's disease (PD) is the association of tremor, rigidity, akinesia-bradykinesia and loss of postural reflexes. Non-motor symptoms such as cognitive impairment may also develop. Frailty is a syndrome characterized by a decrease in physiological reserve that results in an individual's increased vulnerability, which can lead to a variety of adverse factors when exposed to stressors. There are three prominent theoretical frameworks for the study of frailty, the physical model developed by Fried et al., the deficit accumulation model by Rockwood et al. and the biopsychosocial model by Gobbens et al. PD and frailty are highly prevalent in older people and are associated with increased morbidity and mortality. Frailty is a reversible condition, especially during the early stages, so early detection is important. Previous studies have been carried out with the application of exercise programs to reverse frailty in older adults, obtaining good results at a physical level.

General objective:

- Evaluate the effects of a therapeutic home exercise program applied in patients with PD to reverse frailty.

Specific objectives:

* Evaluate the effects of a home therapeutic exercise program on motor and non-motor symptoms, as well as on quality of life, balance and gait.
* Identify the characteristics of the patients who obtain the greatest improvement.
* Evaluate the effects of a home therapeutic exercise program after a period of time of three months after the intervention.

Study design: experimental, prospective, randomized and single-blinded.

Study population: The subjects that will be part of this study will be men and women with a diagnosis of PD belonging to the Health Area V of the Health Service of the Principality of Asturias, Spain.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 60 years or older, with a diagnosis of PD
* Having frailty or prefrailty according to the Fried scale (1 or 2 prefrailty criteria, 3 or more frailty criteria).
* Stage 1-3 of the Hoehn and Yahr scale.
* Patients who have been referred to the Home Rehabilitation Service of the Instituto de Rehabilitación Astur S.A.
* Obtaining a score higher than 24 points in the Mini Mental State Examination (MMSE).
* Signing the informed consent form.

Exclusion Criteria:

* Parkinsonisms secondary, plus or atypical (progressive supranuclear palsy, multiple system atrophy, corticobasal degeneration, Lewy body disease).
* Acute disease causing clinical instability.
* Stage 4 and 5 of the Hoehn and Yahr scale.
* Receiving individualized outpatient or home physiotherapy treatment for Parkinson's disease or secondary parkinsonism.
* Patients unable to speak.
* Patients in terminal phase.
* Patient with dementia.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Frailty: Fried's Frailty Phenotype: | Change in frailty of individuals at baseline up to the 8th and 12th week after interventions.
  Fried's Frailty Phenotype proposed in the Cardiovascular Health Study (Fried et al., 2001) consists of 5 criteria: unintentional weight loss, exhaustion, low physical activity, reduced grip strength, and reduced gait speed. It has a total score ranging from 0 to 5. A frail person is who scores 3 to 5; prefrail when scores 1 to 2, and robust when scores 0.
Frailty: Clinical Frailty Scale. | Change in frailty of individuals at baseline up to the 8th and 12th week after interventions.
  The Clinical Frailty Scale (CFS) was proposed in the Canadian Study of Health and Aging (CSHA) (Rockwood et al., 2005). It is a hierarchical scale of 9 levels ranging from 1, the best state of health, to 9, the worst situation: fit, well, well managed, vulnerable, mildly frail, moderately frail, severely frail, very severely frail, terminally ill.

SECONDARY OUTCOMES:
Comorbidities Charlson Index | Baseline - 8 weeks - 3 months
  It is evaluated according to the Charlson comorbidity index (Charlson et al., 1987). This scale consists of 19 items. Absence of comorbidity between 0 and 1 points, low comorbidity 2 points, high comorbidity between 3 and 5 points and severe comorbidity more than 5 points is considered.
Movement Disorder Society Unified Parkinson´s Disease Rating Scale (MDS-UPDRS). | Baseline - 8 weeks - 3 months
  This tool allows to study the symptoms and the evolution of the disease (Goetz et al., 2008). It is a scale that is subdivided into 4 parts. Part I: non-motor experiences of daily life, comprising 13 items; Part II: motor experiences of daily life, comprising 13 items; Part III: motor exploration, covering 18 items; and Part IV: motor complications, including 6 items. Each question is evaluated from 0 to 4, where 0 is normal and 4 the greater severity, the higher the score the greater involvement (greater impact of PD symptoms).
Cognitive function: Parkinson's Disease Cognitive Rating Scale (PD-CRS). | Baseline - 8 weeks - 3 months
  Parkinson's Disease Cognitive Rating Scale (PD-CRS): It is a scale designed to detect the entire spectrum of cognitive dysfunction that occurs in the course of PD (Pagonabarraga J et al., 2008). It consists of nine cognitive tasks distributed in two sub-scores, with a maximum score of 134 points: fronto-subcortical (fixation verbal memory 12 points, maintained attention 10 points, working memory 10 points, drawing a clock 10 points, deferred verbal memory 12 points, alternating verbal fluence 20 points, action verbal fluence 30 points) and posterior cortical (denomination by confrontation 20 points and copy of a clock 10 points).
Quality of life, PDQ-39 | Baseline - 8 weeks - 3 months
  The Spanish version of the questionnaire Parkinson s disease quality of life questionnaire (PDQ39) is used (Martínez Martín P, et al., 1999, Martínez-Martín P et al., 1998). It consists of 39 items with 5 possible answers. 8 dimensions are analyzed: mobility, daily life activities, emotional well-being, stigma, social support, cognitive impairment, communication and body discomfort. The higher the score, the greater the impact on quality of life.
Short Physical Performance Battery activity level | Baseline - 8 weeks - 3 months
  Physical performance is measured using the Brief Physical Performance Battery (Guralnik et al., 1994). This measure consists of walking 4 m, a balance test with 3 levels (tandem, semi-tandem and feet together) and sitting and reaching 5 times as fast as possible. Total scores range from 0 to 12, with higher scores denoting higher physical performance.
Barthel Index | Baseline - 8 weeks - 3 months
  Functional independence is measured using the Barthel index. It has a total score ranging from 0 to 100, where 0 is the minimum (worst outcome) and 100 is the maximum (best outcome). (Mahoney et al. 1965, Granger et al., 1979).
Lawton Brody Index | Baseline - 8 weeks - 3 months
  Functional independence is measured with the Lawton and Brody Questionnaire (Lawton and Brody, 1969, Vergara I et al., 2012). Instrumental activities of daily living assesses the ability to use the telephone, shop, use transport, cook, do household chores, take medication and manage finances. It has a total score ranging from 0 to 8, with 0 indicating total dependence and the maximum score indicating total independence.
Walking evaluation FAC | Baseline - 8 weeks - 3 months
  It is measured according to the Holden Ambulation Classification (FAC) (Holden et al., 1984). It consists of 6 response categories, from the value 0 (no gear) to the value 5 (independent gear including up and down stairs).
Timed Up and Go (TUG) | Baseline - 8 weeks - 3 months
  Assesses balance, walking difficulties and decreased strength in lower limbs (Poisadlo D and Richardson S, 1991). This test consists of asking the person to get up from a chair with armrests, walk 3 meters, back and sit again, timing the time spent. 10 seconds or less: correct time. Between 10 and 20 seconds: frail marker. Between 20 and 30 seconds risk of falling. More than 30 seconds: high risk of falls.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cruz Sousa Fraguas, Principal Investigator — University of Oviedo
Locations (1):
- University of Oviedo, Oviedo, Spain

REFERENCES:
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Gobbens RJ, van Assen MA, Luijkx KG, Wijnen-Sponselee MT, Schols JM. The Tilburg Frailty Indicator: psychometric properties. J Am Med Dir Assoc. 2010 Jun;11(5):344-55. doi: 10.1016/j.jamda.2009.11.003. Epub 2010 May 8. PMID 20511102
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Martinez-Martin P, Frades Payo B. Quality of life in Parkinson's disease: validation study of the PDQ-39 Spanish version. The Grupo Centro for Study of Movement Disorders. J Neurol. 1998 May;245 Suppl 1:S34-8. doi: 10.1007/pl00007737. PMID 9617722
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Pagonabarraga J, Kulisevsky J, Llebaria G, Garcia-Sanchez C, Pascual-Sedano B, Gironell A. Parkinson's disease-cognitive rating scale: a new cognitive scale specific for Parkinson's disease. Mov Disord. 2008 May 15;23(7):998-1005. doi: 10.1002/mds.22007. PMID 18381647
- [Background] Granger CV, Albrecht GL, Hamilton BB. Outcome of comprehensive medical rehabilitation: measurement by PULSES profile and the Barthel Index. Arch Phys Med Rehabil. 1979 Apr;60(4):145-54. PMID 157729
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Holden MK, Gill KM, Magliozzi MR, Nathan J, Piehl-Baker L. Clinical gait assessment in the neurologically impaired. Reliability and meaningfulness. Phys Ther. 1984 Jan;64(1):35-40. doi: 10.1093/ptj/64.1.35. PMID 6691052
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Qutubuddin AA, Pegg PO, Cifu DX, Brown R, McNamee S, Carne W. Validating the Berg Balance Scale for patients with Parkinson's disease: a key to rehabilitation evaluation. Arch Phys Med Rehabil. 2005 Apr;86(4):789-92. doi: 10.1016/j.apmr.2004.11.005. PMID 15827933
- [Result] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156